CLINICAL TRIAL: NCT04786600
Title: A Phase II Randomized Therapeutic Optimization Trial for Subjects With Refractory Metastatic Colorectal Cancer Using ctDNA: Rapid 1 Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Florida (Other)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF-STO-GI-012; UF-STO-GI-012 (Other: University of Florida); IRB202100341 (Other: University of Florida); OCR40199 (Other: University of Florida)
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; precision oncology; personalized medicine; ctDNA
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Combinations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ctDNA assay-guided intervention (Experimental): Subjects on this arm will be tested with the Signatera ctDNA assay while receiving treatment on a pre-specified sequence of FDA-approved drugs and drug combinations. Subjects will move through this sequence based on the results of the ctDNA assay. Subjects will move to a new drug or drug combination in the sequence when the ctDNA assay indicates a significant increase in ctDNA level. Subjects will also have imaging scans every 12 weeks while on each drug or drug combination and subjects will move to a new drug or drug combination if these scans indicate disease progression.
  Interventions: Device: Signatera ctDNA assay; Drug: pre-specified sequence of FDA-approved drugs and drug combinations
- Scan-guided Intervention (Active Comparator): Subjects on this arm will be treated with the same pre-specified sequence of FDA-approved drugs and drug combinations as those on the ctDNA assay- guided intervention arm. Subjects will move through the sequence based on the results of imaging scans, moving to a new drug or drug combination if imaging shows progressive disease.
  Interventions: Drug: pre-specified sequence of FDA-approved drugs and drug combinations

INTERVENTIONS:
Device: Signatera ctDNA assay — Subjects will be tested with the Signatera ctDNA assay every 2 weeks.
  Arms: ctDNA assay-guided intervention
Drug: pre-specified sequence of FDA-approved drugs and drug combinations — Subjects will receive treatment with a pre-specified sequence of FDA-approved drugs and drug combinations

SUMMARY:
This randomized, phase 2 study will investigate the use of the Signatera ctDNA assay versus the standard scan-based approach to guide treatment in patients with metastatic colorectal cancer. The aim of this study will be to measure and compare the overall survival, progression-free survival, and best overall response while on study of patients whose treatment has been guided by these two approaches.

ELIGIBILITY:
Inclusion Criteria:

* A histologic confirmed adenocarcinoma of the colon or rectum with RECIST measurable metastatic disease measurable and not currently a candidate for oligometastatic definitive management
* Must have at least received first-line oxaliplatin-based therapy for metastatic disease, or a clinically acceptable and documented reason they did not, and progressed or were intolerant to the therapy. Individuals who recurred within 6 months of completion of oxaliplatin based adjuvant chemotherapy are also eligible. Subjects may enroll at any line of therapy past this first line so long as the patient's next clinically reasonable prescribed treatment would be Folfiri + Bevacizumab/biosimilar, Anti-EGFR therapy (with or without irinotecan), OR Lonsurf.
* Subjects must have tissue from either the primary and/or metastatic deposit available for submission at enrollment. Tissue can be from either a biopsy or resection surgery, whichever is most recent, but must be from the past five years.
* Subjects must have tissue and blood shipped to Natera no fewer than 10 days prior to starting treatment.
* Subjects must have had molecular profiling to determine tumor RAS, BRAF and MMR/MSI status
* Subjects with known or suspected Gilbert's disease must be formally tested for UGT1A1*28 with results available to study team prior to treatment initiation
* Any clinically relevant (as deemed by the PI) adverse events related to prior therapies must have resolved to Grade 1 or less (CTCAE 5.0) at study enrollment
* Age ≥18 years
* ECOG performance status of 0-2
* Life expectancy of at least 6 months
* Adequate organ function, as defined as:

  * Absolute neutrophil count (ANC) ≥ 1,500/µL
  * Hemoglobin ≥ 9g/dL
  * Platelets ≥ 100,000/µL
  * Total bilirubin ≤ 1.5 ULN or direct bilirubin ≤ 1 x ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN; if liver metastases present, then AST and ALT must be ≤ 5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 59 mL/min/1.73m using Cockcroft-Gault equation
* Subjects must not have more than one active malignancy at the time of enrollment (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician and approved by the PI] may be included).
* Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 12 weeks after the end of protocol-specified treatment to minimize the risk of pregnancy.
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods throughout the study and should avoid conceiving children for 12 weeks following the last dose of the protocol-specified treatment.
* Written informed consent obtained from the subject and the subject agrees to comply with all the study related procedures

Exclusion Criteria:

* Colorectal cancer known to be Microsatellite High (MSI-H), deficient in DNA mismatch repair genes (dMMR), or BRAF (V600E) mutated
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 12 weeks after the last dose of the protocol-specified treatment
* Females who are pregnant or breastfeeding
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness
* Prior radiation therapy must have been completed 14 days prior to study entry
* Prior chemotherapy or biologic therapy must have been completed 21 days prior to study entry
* Known Dihydropyrimidine Dehydrogenase (DPD) deficiency

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherise Rogers, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm Not Assigned: Subjects in this group were not assigned to an arm due to withdrawing from the study before they could be randomized.
Period: Overall Study
Arm/Group | ctDNA Assay-guided Intervention | Scan-guided Intervention | Arm Not Assigned
Started | 1 | 3 | 2
Completed | 1 | 3 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm Not Assigned: Subjects in this group were not assigned to an arm due to going on study, but were not randomized to either protocol arm due to withdrawal from the study prior to randomization.
- Total: Total of all reporting groups
Arm/Group | ctDNA Assay-guided Intervention | Scan-guided Intervention | Arm Not Assigned | Total
Number analyzed (Participants) | 1 | 3 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 5
  >=65 years | 0 | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 47 [47 to 47] | 63 [55 to 69] | 55.5 [53 to 58] | 57.83 [47 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 1 | 2 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 0 | 2 | 1 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Determine the overall survival
Time Frame: 580 days
Measure: Count of Participants; unit: Participants
Arm/Group | ctDNA Assay-guided Intervention | Scan-guided Intervention
Number analyzed (Participants) | 1 | 3
Participants | 0 | 0

2. Secondary Outcome: Best Overall Treatment Response
Description: Compare the proportion of subjects who receive ctDNA-guided treatment and scan-guided treatment that achieve each RECIST v1.1 response category (complete response, partial response, stable disease, and progressive disease) as their best response while on study treatment. Complete response is defined as the disappearance of all target lesions (any pathological lymph nodes must have reduction in short axis to <10 mm). Partial response is defined as least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of 1 or more new lesions is also considered progression. Stable disease is defined as either sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | ctDNA Assay-guided Intervention | Scan-guided Intervention
Number analyzed (Participants) | 1 | 3
Participants
  Progressive disease | 1 | 3
  Stable disease | 0 | 0
  Partial response | 0 | 0
  Complete response | 0 | 0

3. Secondary Outcome: Progression-free Survival
Description: Determine progression-free survival
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ctDNA Assay-guided Intervention | Scan-guided Intervention
Number analyzed (Participants) | 1 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of randomization until 30 days after the last study visit. Adverse event data were collected for a maximum of 580 days.
Description: Adverse events were assessed by the principal investigator, the treating sub-investigator, and/or the study coordinator from the date of randomization until 30 days after the last study visit. Adverse events were assessed by physical examination, labs, and subject self-reports. Adverse events are not reported for subjects in the "Arm Not Assigned" group because adverse events were only collected for randomized subjects from the date of randomization until 30 days after the last study visit.
Arm/Group | ctDNA Assay-guided Intervention | Scan-guided Intervention
All-Cause Mortality (participants affected / at risk) | 1/1 | 3/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/3
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ctDNA Assay-guided Intervention (N=1) | Scan-guided Intervention (N=3)
Abdominal infection (Infections and infestations) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ctDNA Assay-guided Intervention (N=1) | Scan-guided Intervention (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Decreased absolute basophils (Blood and lymphatic system disorders) | 0 | 1
Decreased C02 total (Blood and lymphatic system disorders) | 0 | 1
Decreased eosinophils (Blood and lymphatic system disorders) | 0 | 1
Increased serum chloride (Blood and lymphatic system disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Creatinine increased (Investigations) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 3
Fever (General disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INR increased (Investigations) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 2
Lymphopenia (Investigations) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Platelet count decreased (Investigations) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 2
Skin infection (Infections and infestations) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
White blood cell decreased (Investigations) | 0 | 3
Weight loss (Investigations) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0
Edema limbs (General disorders) | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT04786600/Prot_SAP_000.pdf